CLINICAL TRIAL: NCT04317040
Title: A Randomized, Double-blind, Placebo-controlled, Multi-site, Phase III Study to Evaluate the Safety and Efficacy of CD24Fc in COVID-19 Treatment
Brief Title: Efprezimod Alfa (CD24Fc, MK-7110) as a Non-antiviral Immunomodulator in COVID-19 Treatment (MK-7110-007)
Acronym: SAC-COVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oncoimmune, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7110-007; 20200674 (Other: WIRB); CD24Fc-007-US (Other: OncoImmune); MK-7110-007 (Other: Merck)
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — CD24 protein, human; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efprezimod alfa (Experimental): Participants receive single dose of 480 mg efprezimod alfa, diluted to 100 ml with normal saline, intravenous (IV) infusion in 60 minutes on Day 1.
  Interventions: Drug: Efprezimod alfa
- Placebo (Placebo Comparator): Participants receive single dose of placebo as normal saline solution 100 ml, IV infusion in 60 minutes, on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efprezimod alfa — Efprezimod alfa is given on Day 1.
  Other Names: Human CD24; Human IgG Fc Fusion Protein; MK-7110
  Arms: Efprezimod alfa
Drug: Placebo — Placebo is given on Day 1.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of efprezimod alfa in hospitalized adult participants who are diagnosed with coronavirus disease 2019 (COVID-19) and receiving oxygen support.

The primary hypothesis of the study is clinical improvement in the experimental group versus the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with coronavirus disease 2019 (COVID-19) and confirmed severe acute respiratory syndrome coronavirus 2 (SARS-coV-2) viral infection
* Severe or critical COVID-19, or National Institute of Allergy and Infectious Diseases (NIAID) 8-point ordinal score 2, 3 or 4 (Scale 2: requiring invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); Scale 3: non-invasive ventilation or high flow oxygen devices; Scale 4: supplemental oxygen support; a peripheral capillary oxygen saturation (SpO2) </= 94% or tachypnea (respiratory rate >/= 24 breaths/min). Intubation should be within 7 days

Exclusion Criteria:

* Participants who are pregnant, breastfeeding, or have a positive pregnancy test result before enrollment
* Participants previously enrolled in the efprezimod alfa study
* Intubation for invasive mechanical ventilation is over 7 days
* Documented acute renal or hepatic failure
* The investigator believes that participating in the trial is not in the best interests of the participant, or the investigator considers unsuitable for enrollment (such as unpredictable risks or subject compliance issues)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (10):
- United States (10):
  - Baptist Health Research Institute, Jacksonville, Florida
  - Anne Anundel Medical Center, Annapolis, Maryland
  - Institute of Human Virology, University of Maryland Baltimore, Baltimore, Maryland
  - Shady Grove Medical Center, Rockville, Maryland
  - White Oak Medical Center, Silver Spring, Maryland
  - Cooper University Hospital, Camden, New Jersey
  - Atlantic Health System, Morristown, New Jersey
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Texas at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Chen GY, Brown NK, Zheng P, Liu Y. Siglec-G/10 in self-nonself discrimination of innate and adaptive immunity. Glycobiology. 2014 Sep;24(9):800-6. doi: 10.1093/glycob/cwu068. Epub 2014 Jul 4. PMID 24996822
- [Background] Liu Y, Chen GY, Zheng P. Sialoside-based pattern recognitions discriminating infections from tissue injuries. Curr Opin Immunol. 2011 Feb;23(1):41-5. doi: 10.1016/j.coi.2010.10.004. Epub 2011 Jan 3. PMID 21208791
- [Background] Chen GY, Chen X, King S, Cavassani KA, Cheng J, Zheng X, Cao H, Yu H, Qu J, Fang D, Wu W, Bai XF, Liu JQ, Woodiga SA, Chen C, Sun L, Hogaboam CM, Kunkel SL, Zheng P, Liu Y. Amelioration of sepsis by inhibiting sialidase-mediated disruption of the CD24-SiglecG interaction. Nat Biotechnol. 2011 May;29(5):428-35. doi: 10.1038/nbt.1846. Epub 2011 Apr 10. PMID 21478876
- [Background] Chen GY, Tang J, Zheng P, Liu Y. CD24 and Siglec-10 selectively repress tissue damage-induced immune responses. Science. 2009 Mar 27;323(5922):1722-5. doi: 10.1126/science.1168988. Epub 2009 Mar 5. PMID 19264983
- [Background] Tian RR, Zhang MX, Zhang LT, Zhang P, Ma JP, Liu M, Devenport M, Zheng P, Zhang XL, Lian XD, Ye M, Zheng HY, Pang W, Zhang GH, Zhang LG, Liu Y, Zheng YT. CD24 and Fc fusion protein protects SIVmac239-infected Chinese rhesus macaque against progression to AIDS. Antiviral Res. 2018 Sep;157:9-17. doi: 10.1016/j.antiviral.2018.07.004. Epub 2018 Jul 3. PMID 29983395
- [Background] Tian RR, Zhang MX, Liu M, Fang X, Li D, Zhang L, Zheng P, Zheng YT, Liu Y. CD24Fc protects against viral pneumonia in simian immunodeficiency virus-infected Chinese rhesus monkeys. Cell Mol Immunol. 2020 Aug;17(8):887-888. doi: 10.1038/s41423-020-0452-5. Epub 2020 May 7. No abstract available. PMID 32382131
- [Derived] Welker J, Pulido JD, Catanzaro AT, Malvestutto CD, Li Z, Cohen JB, Whitman ED, Byrne D, Giddings OK, Lake JE, Chua JV, Li E, Chen J, Zhou X, He K, Gates D, Kaur A, Chen J, Chou HY, Devenport M, Touomou R, Kottilil S, Liu Y, Zheng P; SAC-COVID Study Team. Efficacy and safety of CD24Fc in hospitalised patients with COVID-19: a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Infect Dis. 2022 May;22(5):611-621. doi: 10.1016/S1473-3099(22)00058-5. Epub 2022 Mar 11. PMID 35286843
- [Derived] Song NJ, Allen C, Vilgelm AE, Riesenberg BP, Weller KP, Reynolds K, Chakravarthy KB, Kumar A, Khatiwada A, Sun Z, Ma A, Chang Y, Yusuf M, Li A, Zeng C, Evans JP, Bucci D, Gunasena M, Xu M, Liyanage NPM, Bolyard C, Velegraki M, Liu SL, Ma Q, Devenport M, Liu Y, Zheng P, Malvestutto CD, Chung D, Li Z. Treatment with soluble CD24 attenuates COVID-19-associated systemic immunopathology. J Hematol Oncol. 2022 Jan 10;15(1):5. doi: 10.1186/s13045-021-01222-y. PMID 35012610
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 234 participants enrolled or randomized in the study, 229 participants received study medication and were evaluable for safety analyses.
Groups:
- CD24Fc: Participants received single dose of CD24Fc 480 mg, diluted to 100 ml with normal saline, intravenous (IV) infusion in 60 minutes on Day 1.
- Placebo: Participants received single dose of placebo as normal saline solution 100 ml, IV infusion in 60 minutes on Day 1.
Period: Overall Study
Arm/Group | CD24Fc | Placebo
Started | 116 | 118
Treated | 114 | 115
Completed | 98 | 98
Not Completed | 18 | 20
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 16 | 18
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Incomplete assessments | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | CD24Fc | Placebo | Total
Number analyzed (Participants) | 116 | 118 | 234
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (14) | 57.8 (14.2) | 57.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 89
  Male | 71 | 74 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 44 | 85
  Not Hispanic or Latino | 75 | 74 | 149
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 22 | 50
  White | 53 | 58 | 111
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Time to Improvement in Coronavirus Disease 2019 (COVID-19) Clinical Status
Description: Time to improvement in COVID-19 clinical status: defined as time (days) required from start of treatment to improvement of clinical status severe - moderate/mild or improvement from score 2-4 to ≥5 sustained without drop below 5 within 28 days from randomization, total follow-up period 29 days (Randomization Day 1 + 28 days follow up) per National Institute of Allergy & Infectious Diseases (NIAID) ordinal scale graded: 1=Death; 2=Hospitalized, on invasive mechanical ventilation (IMV)/extracorporeal membrane oxygenation (ECMO); 3=Hospitalized, on non-invasive ventilation (NIV)/high flow oxygen devices; 4=Hospitalized, require supplemental oxygen; 5=Hospitalized, no supplemental oxygen, require medical care; 6=Hospitalized, no supplemental oxygen, don't require medical care; 7=Not hospitalized, limitation on activities &/or require home oxygen; 8=Not hospitalized, no limitations on activities. Median time & 95% confidence intervals (CIs) were reported using Brookmeyer-Crowley method.
Time Frame: Up to Day 29
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 116 | 118
Days | 6.0 [5.0 to 9.0] | 10.5 [7.0 to 15.0]
Statistical Analysis 1: Comparison: CD24Fc vs Placebo; Test type: Other — Hazard ratio (HR) and the associated 95% CIs were calculated based on Cox Regression model and p-value was calculated based on log-rank test, in accordance with the statistical analysis plan; p = 0.0367, Log Rank; Hazard Ratio (HR) = 1.398, 95% CI 2-sided [1.020 to 1.918] — Cox-Regression Model

2. Primary Outcome: Number of Participants Who Experience an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Per protocol, only AEs with Common Terminology Criteria for AE (CTACAE) grade ≥3 were included. The number of participants who experienced an AE were reported.
Time Frame: Up to 30 days
Population: All randomized participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 114 | 115
Participants | 32 | 35

3. Secondary Outcome: Percentage of Participants Who Died or Had Respiratory Failure (RF)
Description: RF was defined as the need for any of the following: 1) mechanical ventilation (MV), 2) ECMO, 3) NIV, or 4) high flow oxygen devices. Percentage of participants who died or had respiratory failure by Day 29 were reported.
Time Frame: Up to Day 29
Population: All randomized participants
Measure: Number; unit: Percentage of Participants
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 116 | 118
Percentage of Participants | 22.4 | 28.0
Statistical Analysis 1: Comparison: CD24Fc vs Placebo; Test type: Other — Risk difference (RD) and the associated 95% CIs were calculated based on Mantel-Haenszel method and p-value was calculated based on Chi-squared test, in accordance with the statistical analysis plan; p = 0.3281, Chi-squared; Risk Difference (RD) = -0.0555, 95% CI 2-sided [-0.1665 to 0.0555] — Mantel-Haenszel method

4. Secondary Outcome: Time to Disease Progression in Clinical Status of COVID-19
Description: Time to disease progression in clinical status is defined as the time (days) for progression from NIAID score (3 or 4) to (2 or 1) or from 2 to 1 within 28 days from randomization, total follow-up period 29 days (Randomization Day 1 + 28 days follow up). NIAID ordinal scale graded as: 1=Death; 2=Hospitalized, on IMV/ECMO; 3=Hospitalized, on NIV/high flow oxygen devices; 4= Hospitalized, require supplemental oxygen; 5=Hospitalized, no supplemental oxygen, require medical care; 6=Hospitalized, no supplemental oxygen, do not require medical care; 7=Not Hospitalized, limitation on activities and/or require home oxygen; 8=Not hospitalized, no limitations on activities.
Time Frame: Up to Day 29
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 116 | 118
Days | NA [NA to NA] — NA = Median, lower and upper limit of 95% CIs for time to disease progression in clinical status of COVID-19 was not reportable at the time of last disease assessment due to insufficient number of participants with events. | NA [NA to NA] — NA = Median, lower and upper limit of 95% CIs for time to disease progression in clinical status of COVID-19 was not reportable at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: CD24Fc vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0306, Log Rank; Hazard Ratio (HR) = 0.558, 95% CI 2-sided [0.327 to 0.954] — Cox Regression Model

5. Secondary Outcome: Number of Participants Who Died Due to Any Cause
Description: Number of participants who died due to any cause were assessed per protocol on Day 15 and Day 29.
Time Frame: Up to Day 29
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 116 | 118
Participants
  Day 15 | 11 | 8
  Day 29 | 16 | 18
Statistical Analysis 1: Comparison: CD24Fc vs Placebo; Day 15; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.4491, Chi-squared; Risk Difference (RD) = 0.0270, 95% CI 2-sided [-0.0430 to 0.0970] — Mantel-Haenszel method used to report all-cause mortality by Day 15
Statistical Analysis 2: Comparison: CD24Fc vs Placebo; Day 29; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.7512, Chi-squared; Risk Difference (RD) = -0.0146, 95% CI 2-sided [-0.1049 to 0.0756] — Mantel-Haenszel method used to report all-cause mortality by Day 29

6. Secondary Outcome: Rate of Clinical Relapse
Description: Rate of clinical relapse was defined as the percentage of participants who had initially reached score 5 on NIAID ordinal scale for more than one day but subsequently became dependent on oxygen support for more than 1 day within 28 days from randomization after initial recovery with a total follow-up period of 29 days (Day 1 of randomization plus 28 days of follow-up). NIAID ordinal scale graded as: 1=Death; 2=Hospitalized, on IMV/ECMO; 3=Hospitalized, on NIV/high flow oxygen devices; 4= Hospitalized, require supplemental oxygen; 5=Hospitalized, no supplemental oxygen, require medical care; 6=Hospitalized, no supplemental oxygen, do not require medical care; 7=Not hospitalized, limitation on activities and/or require home oxygen; 8=Not hospitalized, no limitations on activities. Clopper-Pearson method was used to report the 95% CI.
Time Frame: Up to Day 29
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 116 | 118
Percentage of Participants | 4.3 [1.41 to 9.77] | 6.8 [2.97 to 12.92]

7. Secondary Outcome: Conversion Rate of COVID-19 Clinical Status
Description: Conversion rate of COVID-19 clinical status on days 8 and 15 was defined as the percentage of participants who changed from NIAID ordinal score 2, 3, 4 to score 5 or higher and reported. NIAID ordinal scale graded as: 1=Death; 2=Hospitalized, on IMV/ECMO; 3=Hospitalized, on NIV/high flow oxygen devices; 4= Hospitalized, require supplemental oxygen; 5=Hospitalized, no supplemental oxygen, require medical care; 6=Hospitalized, no supplemental oxygen, do not require medical care; 7=Not hospitalized, limitation on activities and/or require home oxygen; 8=Not hospitalized, no limitations on activities.
Time Frame: Up to Day 15
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 116 | 118
Percentage of participants
  Day 8 | 55.2 [45.7 to 64.4] | 42.4 [33.3 to 51.8]
  Day 15 | 71.6 [62.4 to 79.5] | 55.9 [46.5 to 65.1]

8. Secondary Outcome: Time to Hospital Discharge
Description: The hospital discharge time was defined as the time from randomization to discharge from the hospital and reported. Time to Hospital Discharge (days) from randomization is calculated as: Time to hospital discharge = Date of hospital discharge - Date of randomization.
Time Frame: Up to Day 29
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 116 | 118
Days | 7.0 [6.0 to 9.0] | 10.5 [7.0 to 15.0]
Statistical Analysis 1: Comparison: CD24Fc vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0311, Log Rank; Hazard Ratio (HR) = 1.416, 95% CI 2-sided [1.031 to 1.945] — Cox Regression model

9. Secondary Outcome: Duration of MV
Description: MV included IMV and NIV. Duration of MV (days) was calculated as: End Date of MV - Start Date of MV + 1 and reported.
Time Frame: Up to Day 29
Population: All randomized participants who received MV
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 28 | 39
Days | 14.3 (12.34) | 14.3 (8.85)

10. Secondary Outcome: Duration of Pressors
Description: Pressor administration included norepinephrine, epinephrine, vasopressin, dopamine and phenylephrine. Duration of pressor (days) was defined as: End Date of Pressor - Start Date of Pressor + 1 and reported.
Time Frame: Up to Day 29
Population: All randomized participants who received pressors
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 20 | 24
Days | 6.3 (5.59) | 7.9 (8.86)

11. Secondary Outcome: Duration of ECMO
Description: Duration of ECMO treatment (days) was calculated as: End Date of ECMO Treatment - Start Date of ECMO Treatment + 1 and reported.
Time Frame: Up to Day 29
Population: All randomized participants who received ECMO
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 0 | 1
Days |  | 11.0 (NA) — NA = Standard deviation for duration of ECMO treatment was not reportable at the time of last disease assessment due to insufficient number of participants with events.

12. Secondary Outcome: Duration of High Flow Oxygen Therapy
Description: Duration of oxygen therapy (oxygen inhalation by high flow nasal cannula or mask) (days) was calculated as: End Date of high flow oxygen therapy - Start Date of high flow oxygen therapy + 1 and reported.
Time Frame: Up to Day 29
Population: All randomized participants who received high flow oxygen therapy
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 114 | 115
Days | 13.8 (12.91) | 13.0 (10.12)

13. Secondary Outcome: Length of Hospital Stay
Description: Length of Hospital Stay (Days) was defined as date of discharge - date of admission + 1 and reported. Data presented below include hospitalization time prior to enrollment in the study with total duration of up to 90 days.
Time Frame: Up to 90 days
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 116 | 118
Days | 16.6 (16.27) | 18.2 (13.54)

14. Secondary Outcome: Change From Baseline in Absolute Lymphocyte Count
Description: Blood samples were collected to present the change from baseline in the absolute lymphocyte count on days 1, 4, 8, and 15 in peripheral blood. To calculate the change from baseline in absolute lymphocyte count at specific timepoints (Days 1, 4, 8 and 15), only the participants who had both, a baseline, and a post baseline value at the specific timepoint (Days 1, 4, 8 and 15) were included in the analysis.
Time Frame: Baseline and up to Day 15
Population: All randomized participants with lymphocyte data available
Measure: Mean (Standard Deviation); unit: 10^9 Cells/Liter
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 114 | 114
10^9 Cells/Liter
  Baseline: number analyzed (Participants) | 113 | 113
  Baseline | 2.357 (5.1173) | 2.437 (4.7660)
  Day 1: number analyzed (Participants) | 30 | 29
  Day 1 | 5.317 (8.0772) | 5.125 (7.3979)
  Day 4: number analyzed (Participants) | 89 | 96
  Day 4 | 2.373 (5.7549) | 2.461 (4.2074)
  Day 8: number analyzed (Participants) | 51 | 61
  Day 8 | 2.557 (4.7147) | 1.839 (2.7319)
  Day 15: number analyzed (Participants) | 23 | 39
  Day 15 | 1.965 (3.8555) | 2.378 (4.6402)
  Change from Baseline to Day 1: number analyzed (Participants) | 30 | 29
  Change from Baseline to Day 1 | 0.374 (2.0467) | -0.148 (0.7985)
  Change from Baseline to Day 4: number analyzed (Participants) | 88 | 95
  Change from Baseline to Day 4 | 0.219 (5.2971) | 0.053 (2.2800)
  Change from Baseline to Day 8: number analyzed (Participants) | 50 | 60
  Change from Baseline to Day 8 | 0.575 (5.5692) | -0.491 (3.1128)
  Change from Baseline to Day 15: number analyzed (Participants) | 22 | 39
  Change from Baseline to Day 15 | 0.558 (4.3613) | -0.280 (5.1603)

15. Secondary Outcome: Change From Baseline in D-Dimer Concentration
Description: Blood samples were collected to present the change from baseline in the D-dimer concentration on days 4, 8 and 15 in peripheral blood. To calculate change from baseline in D-dimer concentration at specific timepoints (Days 4, 8 and 15), only the participants who had both, a baseline, and a post baseline value at the specific timepoint (Days 4, 8 and 15) were included in the analysis.
Time Frame: Baseline and up to Day 15
Population: All randomized participants with D-dimer concentration data available
Measure: Mean (Standard Deviation); unit: nmol/Liter
Arm/Group | CD24Fc | Placebo
Number analyzed (Participants) | 104 | 108
nmol/Liter
  Baseline: number analyzed (Participants) | 102 | 103
  Baseline | 153.717 (1457.6865) | 9.767 (12.4347)
  Day 4: number analyzed (Participants) | 63 | 73
  Day 4 | 10.451 (16.1924) | 13.885 (33.0328)
  Day 8: number analyzed (Participants) | 39 | 52
  Day 8 | 13.224 (17.4246) | 13.349 (17.2777)
  Day 15: number analyzed (Participants) | 18 | 33
  Day 15 | 11.700 (7.9524) | 13.892 (19.9369)
  Change from Baseline to Day 4: number analyzed (Participants) | 61 | 70
  Change from Baseline to Day 4 | -0.427 (9.6796) | 3.971 (34.9427)
  Change from Baseline to Day 8: number analyzed (Participants) | 37 | 49
  Change from Baseline to Day 8 | -397.547 (2419.1594) | 0.703 (18.3254)
  Change from Baseline to Day 15: number analyzed (Participants) | 18 | 29
  Change from Baseline to Day 15 | 3.076 (10.0044) | -3.591 (19.0945)

ADVERSE EVENTS:
Time Frame: Serious adverse events (AEs), non-serious AEs and all-cause mortality were collected up to approximately 30 days.
Description: All-cause mortality was reported on all randomized participants. Serious and non-serious AEs were reported among participants who received at least one dose of study treatment.
Arm/Group | CD24Fc | Placebo
All-Cause Mortality (participants affected / at risk) | 16/116 | 18/118
Serious Adverse Events (participants affected / at risk) | 26/114 | 27/115
Other Adverse Events (participants affected / at risk) | 0/114 | 0/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD24Fc (N=114) | Placebo (N=115)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Pulse absent (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 14 (14)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will support writing and publication of scientific reports, journal papers and oral presentations by the study principal investigator and others making scientific contribution to the research effort. Any reports, papers, and/or presentations must be reviewed and approved prior to submitting for publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT04317040/Prot_SAP_000.pdf